CLINICAL TRIAL: NCT03896061
Title: A Videographic Study to Evaluate the Impact of a Pulsed Firing Technique on Staple Line Interventions in Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC-2018-01
Record Dates: First submitted 2019-03-12; First posted 2019-03-29 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Hemostasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Laparoscopic sleeve procedures — Laparoscopic sleeve procedures with powered stapler

SUMMARY:
Prospective, multi-center study will evaluate a pulsing technique with the ECHELON FLEX GST system for hemostasis at the staple line in laparoscopic sleeve gastrectomy procedures.

DETAILED DESCRIPTION:
Prospective, multi-center study will evaluate a pulsing technique with the ECHELON FLEX GST system for hemostasis at the staple line in laparoscopic sleeve gastrectomy procedures.

Data collected for the study consists of videography imaging and audio. Video recordings (no subject identifiers) will involve the use of two cameras providing:

1. Synchronized Internal and external views of devices used, including the hands of the surgeon firing the endocutter; and
2. Audio of the procedure to record the motor noise of the device while firing (audio will help identify the surgeon's pulsing technique during the procedure).

Surgeon satisfaction with transection technique will also be collected. Videography will be evaluated for staple line hemostasis and need for surgical intervention at the staple line (defined in Criteria for Evaluation).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign a Video, Audio and Digital Data Release consent for participation; and
* Scheduled for a laparoscopic sleeve gastrectomy procedure.

Exclusion Criteria:

* Prophylactic use of buttressing material
* Other staple line reinforcement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who satisfy inclusion/exclusion criteria for informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of oozing/bleeding at the staple line | Intraoperative
  Investigate whether use of a prescribed pulsing technique may provide potential reduction in the occurrence of oozing/bleeding at the staple line.
Occurence of sugical interventions required to achieve hemostasis at the staple line | Intraoperative
  Investigate whether use of a prescribed pulsing technique may provide potential reduction in the occurrence of surgical interventions required to achieve hemostasis at the staple line.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Surgical Specialists of Louisiana, Metairie, Louisiana
  - State University of New York at Buffalo, Buffalo, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu